CLINICAL TRIAL: NCT03729193
Title: Assessment of Musculoskeletal Pain and Psychosocial Status of Athletes in Different Disciplines
Brief Title: Assessment of Musculoskeletal Pain and Psychosocial Status of Athletes
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, amine atac, research assistant, Istanbul Medipol University Hospital
Other Study IDs: 10840098-604.01.01-E.45126
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Pain
Keywords: musculoskeletal system pain; athlete; psychosocial problems; algometer
MeSH Terms: conditions — Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- soccer players: Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of 20 soccer players.
  Interventions: Behavioral: Measuring devices and questionnaires
- basketball players: Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of 20 basketball players.
  Interventions: Behavioral: Measuring devices and questionnaires
- volleyball players: Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of 20 volleyball players.
  Interventions: Behavioral: Measuring devices and questionnaires
- archers: Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of 20 archers.
  Interventions: Behavioral: Measuring devices and questionnaires
- kickboxers: Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of 20 kickboxers.
  Interventions: Behavioral: Measuring devices and questionnaires
- table tennis athletes: Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of 20 table tennis athletes.
  Interventions: Behavioral: Measuring devices and questionnaires
- runners: Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of 20 runners.
  Interventions: Behavioral: Measuring devices and questionnaires
- field tennis athletes: Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of 20 field tennis athletes.
  Interventions: Behavioral: Measuring devices and questionnaires

INTERVENTIONS:
Behavioral: Measuring devices and questionnaires — Measuring devices and questionnaires will be applied to assess the pain and psychosocial states of musculoskeletal system of athletes. The Expanded Scandinavian Muscle Skeleton Questionnaire (NMQ) and Visible Analogue Scale (VAS) will be used to identify and assess the symptoms of musculoskeletal discomfort as 'pain'. The participant will be evaluated with the algometer for identifying their pain threshold, the sporty trust will be questioned with the Sporty Trust Continuous Inventory, and the Quality of Life will be assessed with the World Health Organization Quality of Life Scale Short Form and Depression will be evaluated with Beck Depression Inventory.

SUMMARY:
The sporty performance exhibited by an athlete faces physiological, biomechanical and psychological activity of the athlete. It depends on both the psychological state and the elevation of the musculoskeletal system to a certain level so that the athlete can perform optimally and excellently. For this reason, we aimed to evaluate the musculoskeletal system pain of amateur and professional athletes in different disciplines and the psychosocial states such as sports confidence, depression and quality of life.

DETAILED DESCRIPTION:
This study consists of 160 sportsmen who are participating in sports by doing sports in soccer, basketball, volleyball, athletics, table tennis, field tennis, kickboxing and archery branches between the ages of 15 and 36. The Expanded Scandinavian Muscle Skeleton Questionnaire (NMQ) and Visible Analogue Scale (VAS) will be used to identify and assess the symptoms of musculoskeletal discomfort as 'pain'. The participant will be evaluated with the algometer for identifying their pain threshold, the sporty trust will be questioned with the Sporty Trust Continuous Inventory, and the Quality of Life will be assessed with the World Health Organization Quality of Life Scale Short Form and Depression will be evaluated with Beck Depression Inventory.

ELIGIBILITY:
Inclusion Criteria:

* The athletes and their coaches must be voluntary and willing.
* During the evaluation, the athletes must give careful and relevant answers to the measuring instruments.
* They have to actively run the sport they belong to.
* The dominant upper extremity should be the right side.

Exclusion Criteria:

* Having undergone a surgical operation due to sports injuries in the last 3 weeks
* The athletes do not want to answer the surveying instruments

Ages: 15 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will be between the ages of 15 and 36.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-12-30 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Musculoskeletal system pain | 14 days
  Extended Nordic Musculoskeletal Questionnaire consists of 11 questions asked from the 9 body regions. The questionnaire firstly questions the pain-pain sensation in the 9 body areas in the form of a yes / no response.
severity of pain perception | 14 days
  Visual Analogue Scale (VAS); This study will be used to understand how the athlete expresses pain on a 10 cm scale before, during and after training. Using a ruler, the score is about 10-cm in length. It have been recommended: no pain (0 and4 mm), mild pain (5-44 mm), moderate pain (45 mild74 mm), and severe pain (75 :100 mm). the VAS values of the athletes will be questioned for in the resting, before and after the training.
pain threshold | 14 days
  The pain threshold of the right hand and the left hand will be measured in kilograms (kg) with the algometer. A difference of 2 kg between the measured right and left sides, or less than 3 kg of the measured side, indicates that the pain threshold is low and abnormal.

SECONDARY OUTCOMES:
Sporty confidence | 14 days
  Participants' sporty confidence will asses by using Continuous Sportive Trust ınventory. This sport-specific inventory consists of a 9-point Likert scale which is engaged in 1 (low) and 9 (high) items from 13 items without sub-components. The level of continuous sporty confidence is obtained by the mean score obtained by collecting the scores of 13 items and dividing them by 13. 1-3 points means low level sporting self-confidence, 4-6 points medium level sporting self-confidence, 7-9 points high level sporting self-confidence.
Health Related Quality of Life | 14 days
  Participants' health Related Quality of Lifequality of life will asses by using World Health Organization Quality of Life Scale Short Form (WHOQOL-BREF). This scale consists of 26 questions that measure overall quality of life and overall health. The other 24 questions are divided into four areas: the physical health title consists of 7 questions, the psychological health title consists of 6 questions, the social relationship title is 3 questions and the environmental health title consists of 8 questions.
  Each title is scored independently. Each item is scored on a Likert-type scale from 1 to 5. The scores are then calculated for each quality of life subtitle and converted to 0-100 points. A high score means that the quality of life is high.
Depression | 14 days
  Participants' depression will asses by using Beck Depression Inventory. The Beck Depression Inventory was a 21-item self-drawing questionnaire to measure depressive symptoms in clinical and non-clinical populations for Beck et al. Its substance has 4 possible answers to a Likert-type scale found between 0 (none) and 3 (irresistible). High scores indicate severe depressive symptoms: 0-13 points or minimal depression, 14-19 mild, 20-28 moderate and 29-63 indicate severe depression level.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Şahin, Study Director — Medipol University
Locations (1):
- Istanbul Medipol Universıty, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahraman T, Genc A, Goz E. The Nordic Musculoskeletal Questionnaire: cross-cultural adaptation into Turkish assessing its psychometric properties. Disabil Rehabil. 2016 Oct;38(21):2153-60. doi: 10.3109/09638288.2015.1114034. Epub 2016 Jan 4. PMID 26726840
- [Background] Aghilinejad M, Choobineh AR, Sadeghi Z, Nouri MK, Bahrami Ahmadi A. Prevalence of Musculoskeletal Disorders among Iranian Steel Workers. Iran Red Crescent Med J. 2012 Apr;14(4):198-203. Epub 2012 Apr 1. PMID 22754681
- [Background] Wang YP, Gorenstein C. Psychometric properties of the Beck Depression Inventory-II: a comprehensive review. Braz J Psychiatry. 2013 Oct-Dec;35(4):416-31. doi: 10.1590/1516-4446-2012-1048. Epub 2013 Dec 23. PMID 24402217
- See also: Pubmed link — https://www.ncbi.nlm.nih.gov/pubmed/26726840?dopt=Abstract
- See also: Pubmed link — https://www.ncbi.nlm.nih.gov/pubmed/22754681?dopt=Abstract
- See also: Pubmed link — https://www.ncbi.nlm.nih.gov/pubmed/24402217?dopt=Abstract